CLINICAL TRIAL: NCT07268989
Title: Evaluation of Mechanical Power to Predict Weaning Success in the Intensive Care Unit: A Prospective Observational Study
Brief Title: Evaluation of Mechanical Power and Ventilator Parameters to Predict Weaning Success in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Anıl Berkay Balıtatlı (Other)
Responsible Party: Sponsor-Investigator, Anıl Berkay Balıtatlı, Resident Physician (Anesthesiology and Intensive Care), Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: Mechanical Power
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Weaning Mechanical Ventilation; Mechanical Power; Negative Inspiratory Force; Airway Occlusion Pressure
Keywords: Mechanical power; Weaning mechanical ventilation; Negative inspiratory; Airway occlusion pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated ICU Patients Undergoing Weaning: Adult patients receiving mechanical ventilation in the intensive care unit (ICU) who meet clinical criteria for planned weaning and extubation. All patients will undergo bedside ventilator-based respiratory assessment to evaluate mechanical power (MP), airway occlusion pressure (P0.1), negative inspiratory force (NIF), and the rapid shallow breathing index (RSBI) prior to extubation.
  Interventions: Diagnostic Test: Mechanical power

INTERVENTIONS:
Diagnostic Test: Mechanical power — Non-invasive bedside evaluation of respiratory load, neural drive, and inspiratory muscle capacity using mechanical power (MP), airway occlusion pressure (P0.1), negative inspiratory force (NIF), and the rapid shallow breathing index (RSBI).
  • Measurements will be performed once within 2 hours prior to the extubation decision as part of routine ICU respiratory monitoring.

SUMMARY:
The goal of this prospective observational study is to evaluate whether ventilator-based respiratory parameters can predict weaning success in adult intensive care unit (ICU) patients who are mechanically ventilated. The main questions it aims to answer are:

Can the mechanical power (MP) value predict successful extubation? Do other respiratory parameters-airway occlusion pressure (P0.1), negative inspiratory force (NIF), and the rapid shallow breathing index (RSBI)-provide additional prognostic value for weaning outcomes?

Participants will:

* Be adult ICU patients planned for weaning from mechanical ventilation.
* Undergo bedside ventilatory assessment within 2 hours after meeting clinical weaning criteria.
* Have the following respiratory parameters measured: MP, P0.1, NIF, and RSBI.
* Be monitored for 48 hours after extubation to assess weaning success (defined as no need for reintubation, non-invasive ventilation, or high-flow oxygen support)

DETAILED DESCRIPTION:
This is a prospective, observational, single-center study designed to investigate whether ventilator-derived physiological measurements can predict weaning success in mechanically ventilated adult ICU patients. The primary objective is to determine the prognostic value of mechanical power (MP) in forecasting successful extubation.

Secondary objectives include the evaluation of additional respiratory parameters such as airway occlusion pressure (P0.1), negative inspiratory force (NIF), the rapid shallow breathing index (RSBI), and the mechanical power/negative inspiratory force ratio (MP/NIF). These parameters will be measured at the bedside within 2 hours after patients meet clinical weaning criteria and are hemodynamically stable.

All participants will be monitored for 48 hours after extubation. Weaning success is defined as the ability to sustain spontaneous breathing without the need for reintubation, non-invasive ventilation, or high-flow oxygen therapy during this period.

Data collection will include:

Respiratory measurements obtained from the ventilator: MP, P0.1, NIF, RSBI, and MP/NIF.

Demographic and clinical data: age, sex, BMI, ICU admission diagnosis, APACHE II and SOFA scores, ventilator settings, and duration of mechanical ventilation.

Post-extubation follow-up: reintubation, non-invasive ventilation or high-flow oxygen use, SpO₂ values, blood gas analysis, and vital signs.

This study does not involve any interventions beyond standard ICU care. Ventilator-based respiratory assessments are routinely performed in ICU settings and pose no additional risk to participants.

The results may support the integration of load-drive-capacity assessment into routine ICU weaning protocols and improve clinical decision-making by reducing the incidence of weaning failure and associated complications.

ELIGIBILITY:
Inclusion Criteria:

-

Age ≥ 18 years (adult patient population)

* Patients receiving invasive mechanical ventilation in the intensive care unit
* Having been intubated for at least 24 hours
* Patients for whom the clinical team has decided extubation and who meet the following weaning criteria:
* Stable respiratory parameters (FiO₂ ≤ 40%, PEEP ≤ 5 cmH₂O, SpO₂ ≥ 92%)
* Hemodynamic stability (no inotropic support or minimal/stable dose)
* Appropriate neurological status (able to follow commands)
* Stable acid-base balance
* Adequate secretion control
* Technically suitable ventilator and measurement conditions
* Written informed consent obtained from the patient or legal representative

Exclusion Criteria:

* Patients with any of the following conditions will be excluded:

and

* Individuals under 18 years of age
* Pregnant patients
* Patients who do not meet the weaning criteria
* Tracheostomized patients
* Neuromuscular diseases (e.g., Guillain-Barré syndrome, Duchenne muscular dystrophy, etc.)
* Technical inadequacy preventing correct ventilator measurements
* Significant asynchrony (e.g., auto-PEEP, double triggering, ineffective triggering, cycle asynchrony, auto-triggering)
* Patients without an extubation plan or those receiving palliative care
* RASS ≤ -2 (excessive sedation) for PSV mode measurements
* RASS ≥ +2 (agitation) for PSV-CPAP mode measurements
* Patients with delirium for PSV-CPAP mode measurements
* Patients who cannot provide consent, have no legal representative, or whose representative refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are receiving invasive mechanical ventilation in the intensive care unit (ICU) and are scheduled for planned extubation based on standard clinical weaning criteria. All participants must be hemodynamically stable and able to undergo bedside ventilator-based respiratory assessment, including mechanical power (MP), airway occlusion pressure (P0.1), negative inspiratory force (NIF), and the rapid shallow breathing index (RSBI), prior to extubation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power (MP) | 48 hour
  Mechanical Power (MP), a ventilator-derived estimate of the total mechanical energy transferred to the respiratory system per unit time, will be measured prior to planned extubation and evaluated in relation to extubation outcomes

SECONDARY OUTCOMES:
Airway Occlusion Pressure at 100 ms (P0.1) | 48 hour
  P0.1, an indicator of the patient's neural inspiratory drive that reflects the initial negative pressure generated at the start of a breath, will be measured prior to planned extubation and evaluated in relation to extubation outcomes
Negative Inspiratory Force (NIF) | 48 hour
  NIF, a measure of maximal inspiratory muscle strength reflecting the patient's ability to generate negative pressure, will be obtained prior to planned extubation and evaluated in relation to extubation outcomes
Rapid Shallow Breathing Index (RSBI) | 48 hour
  RSBI, an established index that incorporates respiratory rate and tidal volume to characterize rapid and shallow breathing, will be recorded prior to planned extubation and evaluated in relation to extubation outcomes
Mechanical Power to Negative Inspiratory Force Ratio (MP/NIF Ratio) | 48 hour
  The MP/NIF ratio, reflecting the relationship between ventilatory mechanical load and inspiratory muscle capacity, will be calculated prior to planned extubation and evaluated in relation to extubation outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided